CLINICAL TRIAL: NCT01462019
Title: Photobiomodulation as a New Approach for the Treatment of Nipple Traumas
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pontifícia Universidade Católica de Minas Gerais (Other)
Responsible Party: Principal Investigator, Angelica Rodrigues de Araujo, Profa., Phd, Pontifícia Universidade Católica de Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0239.0.213.000-07
Record Dates: First submitted 2011-10-26; First posted 2011-10-28 (Estimated); Last update posted 2011-10-28 (Estimated); Status verified 2011-10

CONDITIONS: Injuries to the Nipple (Fissures and Cracks) Resulting Breastfeeding
Keywords: nipple trauma; breast feeding; phototherapy; wound healing
MeSH Terms: conditions — Breast Feeding | interventions — Low-Level Light Therapy

ARMS (2):
- Control (No Intervention)
- Photobiomodulation (Experimental)
  Interventions: Device: Photobiomodulation

INTERVENTIONS:
Device: Photobiomodulation — the participants of this group will receive, in addition to guidance on the breast care and proper techniques for feeding, phototherapy applications through photobiomodulador a device developed specifically for the treatment of nipple injuries. The parameters for applications are: continuous mode of emission, power output 10 mW, wavelength infrared (scanning from 880 to 904 nm) fluence of 4 J / cm ² and total application time of 10 minutes.
  The application of the device will be three times per week on alternate days for seven consecutive weeks, totaling 21 sessions.
  Arms: Photobiomodulation

SUMMARY:
Inadequate care during pregnancy and postpartum are predisposing factors for the emergence of nipple fissures. The therapeutic approach of nipple trauma care guidelines aimed at the breast and the appropriate techniques for breastfeeding. These measures, however, have a much more preventive than curative, it is not, in most cases, sufficient to power the closing of nipple trauma. The objective of this study was to evaluate the effectiveness of a phototherapy device designed specifically for the treatment of nipple trauma.

ELIGIBILITY:
Inclusion Criteria:

* women should have a medical diagnosis of nipple trauma were not infected and aged 18 to 35 years

Exclusion Criteria:

* previous history of cancer; use of other therapeutic modalities that might interfere with the healing of the lesions; presence of infected wounds; history of photosensitivity to light; cognitive deficits that undermine the understanding and implementation of guidelines of care for breast

Ages: 18 Years to 35 Years | Sex: Female
Age Groups: Adult
Dates: Start 2006-02; Primary Completion 2006-08 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Size and classification of injuries
  wounds nipple will be measured weekly in the initial assessment and for six consecutive weeks, using a digital caliper and classified at the beginning and end of treatment according to Pereira et al (1998). The measurements and classification of cracks will be conducted by a researcher previously trained to perform procedures.

SECONDARY OUTCOMES:
Pain:
  pain intensity will be evaluated using the Visual Numeric Scale (VNS). The EVN will be applied at baseline and at the beginning of each week of treatment, for six consecutive weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Pontifícia Universidade Católica de Minas Gerais, Belo Horizonte, Minas Gerais, Brazil